CLINICAL TRIAL: NCT03942302
Title: Characterization of Variable MARrcha's Diary Variables as a Useful Measure of Physical Activity in Patients With Physical COPD in Patients With COPD
Brief Title: Characterization of Variable MARrcha's Diary Variables as a Useful Measure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ferran Morell (Other)
Responsible Party: Sponsor-Investigator, Ferran Morell, Director, Fundacio Catalana de Pneumologia
Organization: Fundacio Catalana de Pneumologia (Other)
Other Study IDs: FUC-EPO-2018-01
Record Dates: First submitted 2019-04-15; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validate a simple clinical tool to evaluate physical activity (the question "How many minutes does it walk per day?" Or equivalent), compared to the rest of the collected physical activity data (PROactive questionnaire and objective physical activity data by means of an accelerometer record) in patients with COPD.

DETAILED DESCRIPTION:
Observational, national and multicenter epidemiological study in adult patients with COPD that will take place in the consultations of specialists in pneumology under conditions of usual clinical practice and that will be developed in two visits per patient.

ELIGIBILITY:
Inclusion Criteria:

Adult patients, ≥ 40 years.

* Patients diagnosed with COPD according to the GOLD criteria: FEV1 / FVC postbronchodilator <0.70 in a spirometry performed in the last 12 months.
* Smokers or ex-smokers of ≥10 pack-years.
* Patients with a minimum age in the diagnosis of COPD of at least 6 months.
* Patients who accept their participation in the study and who have given their informed consent (IC) in writing to participate in it.

Exclusion Criteria:

* Patients whose clinical history data are not available.
* Patients unable to understand the study questionnaires.
* Patients with physical limitation (not caused by the respiratory disease, eg disability, orthopedic limitation, etc.) and / or psychic that prevents the proper conduct of the study.
* Patients who present a moderate or severe exacerbation of COPD in the month prior to inclusion.
* Patients with other chronic respiratory diseases other than COPD (such as cystic fibrosis, bronchiectasis of origin other than COPD, neoplasia, pneumonia).
* Patients with serious cardiovascular or neurological diseases.
* Hospital admission for any reason in the month prior to inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population under study will be constituted by adult patients diagnosed with COPD.
  To avoid selection biases, each participating researcher will include in the study the first 10 patients who come to a pulmonology clinic with a clinical diagnosis of COPD and who meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Minutes of daily walking | During the 7 days that the device has.
  For such effects, the level of physical activity will be determined through a unique question, formulated in 5 different ways, which aims to collect the minutes of physical activity or daily walking minutes. The one that best fits the objective of the study will be selected.
  The questions that will be asked will be:
  1. How many minutes do you walk per day, on average?
  2. How many minutes do you walk briskly a day, on average?
  3. How many minutes do you walk outside the home on average?
  4. How many minutes do you spend doing physical activity a day, on average?
  5. How many minutes per day do you engage in moderate to intense physical activity, such as brisk walking, cycling, working in the garden, swimming, dancing, etc., on average?

SECONDARY OUTCOMES:
Date of inclusion in the study | day 9
  [day-month-year]
Age | day 9
  [date of birth, day-month-year]
Sex | day 9
  [male / female]
Size | day 9
  [cm]
Weight | day 9
  [kg]
Body Mass Index | day 9
  (BMI) [kg / m2]
Marital Status | day 9
  [single / married / separated / divorced / widowed]
Family situation | day 9
  Coexistence situation [only (a) / accompanied)
  * Has children? [if not]
  * If yes, how many children? [and ages for each child]
  * Does any child live in the family home? [if not]
  * Number of children in the family home [ages of these children]
  * Do you have grandchildren? [if not]
  * If yes, how many grandchildren? [and ages for each grandchild]
  * Care for your grandchildren on a regular basis? [if not]
  * Age of each grandchild in care
  * Frequency with which she takes care of grandchildren [times / week]
  * Do you have dog / s? [if not. If yes, specify how many]
Place of residence | day 9
  [house / flat / others, specify]
Academic training | day 9
  [without studies, primary, secondary, university studies]
Employment status | day 9
  [self-employed / self-employed / unemployed / retired (a) / household tasks / other, specify]
Socioeconomic level | day 9
  family income 15000€/15000€-25000€/25000€-30000€/>30000€
Smoking | day 9
  [yes / ex]
  * If yes, how many cigarettes / day now? How many packages / year? How many years of current smoking?
  * In the case of an ex-smoker, how many cigarettes / day did he smoke? How many packages / year did he smoke? How many years of previous smoking? How many years / months without smoking until the start of the study?
Date | day 9
  [day-month-year]
Description of instruments and measures | day 9
  Spirometry is a test of lung function (flow and capacity) that evaluates the amount of air through exhalation. The forced spirometry, in particular, is based on making the patient after a maximum inspiration exhale all the air, in the shortest time possible.
  [forced expiratory volume the first second (FEV1) in milliliters / forced vital capacity (FVC) in milliliters / FEV1 / FVC ratio (FEV1%)
FEV1 | day 9
  it is a measure of flow and is expressed in milliliters and is the maximum volume exhaled in the first second of a forced expiration. Its normal value is> 80% of the theoretical value.
FVC | day 9
  it is a measurement of capacity that is expressed in milliliters and is the maximum volume of exhaled air with the maximum possible effort, based on the total volume that the patient expels from maximum inspiration to maximum expiration. Its normal value is> 80% of the theoretical value.
FEV1% | day 9
  it is indicative of the percentage of the total volume expired during the first second. Its normal value is> 70-75% of the theoretical value.
Phenotype of COPD | day 9
  [non-exacerbator / mixed COPD-asthma / exacerbation with emphysema /exacerbator with chronic bronchitis]
Non-pharmacological treatment | day 9
  [smoking cessation / rehabilitation program / oxygen therapy / others, specify]
Number and scope of treatment of exacerbations suffered in the last year | day 9
  [ambulatory / hospital]
Date of the last moderate-severe exacerbation. | day 9
  [day-month-year]
Scales, questionnaires and indexes | day 9
  * IMC
  * FEV1% Dyspnea (from the modified MRC scale)
  * Distance collected in the 6MW [meters]
  * Serious exacerbations in the last 12 months (only visits to hospital emergencies or admissions are included) [number of exacerbations]
  * Determination of the prognostic severity according to BODEX data [three levels: I (mild of 0-2 points), II (moderate, 3-4 points), III (severe, ≥5 points)].
  * COTE comorbidity index, calculated according to 10 comorbidities to be assessed with variable scores, between 1 and 6 points [see Annex 9 for the complete list of comorbidities to be analyzed]
Spirometry | day 9
  * FEV1: is a measure of flow and is expressed in milliliters and is the maximum volume expired in the first second of a forced expiration. Its normal value is> 80% of the theoretical value.
  * FVC: is a measure of capacity that is expressed in milliliters and is the maximum volume of exhaled air with the maximum possible effort, based on the total volume that the patient expels from maximum inspiration to maximum expiration. Its normal value is> 80% of the theoretical value.
  * Ratio FEV1 / FVC x 100 (FEV1%): it is indicative of the percentage of the total expired volume during the first second. Its normal value is> 70-75% of the theoretical value.
BODE and BODEX Index (Annex 8) | day 9
  * The BODE index integrates the BMI, the FEV1, the degree of dyspnea (through the data of the modified MRC scale) and the exercise capacity evaluated by means of a 6-minute walk test. The scores of each variable range from 0 to 3 (range 0-10). An increase in one point of the BODE index is associated with a 34% increase in mortality from all causes and 62% in mortality from respiratory causes.
  * The BODEX index takes into account the number of severe exacerbations (visits to hospital emergencies and admissions) instead of the walking test. The scores for each variable range from 0 to 3 (range 0-9). If the BODEx index is ≥ 5 points, the exercise test will be taken into account to determine the level of severity. Three levels of prognostic severity of COPD will be established: I (mild of 0-2 points), II (moderate, 3-4 points), III (severe, ≥5 points).
COTE comorbidity index (annex 9) | day 9
  The COTE index (Divo et al., 2012) describes 10 comorbidities: cancer (lung, esophagus, pancreas and breast) (6 points), other cancers (2 points), anxiety (in women, 6 points), liver cirrhosis (2 points), atrial fibrillation (2 points), diabetes with neuropathy (2 points), pulmonary fibrosis (2 points), congestive heart failure (1 point), gastroduodenal ulcer (1 point) and coronary disease (1 point) (range) 0-25). A score ≥ 4 increases more than 2 times the expected risk of death.
Charlson comorbidity index (InCC) (Annex 10) | day 9
  The Charlson comorbidity index (Charlson et al., 1987) is a 10-year survival assessment system, depending on the age of the patient being evaluated and the comorbidities of the subject. In addition to age, it consists of 19 items, which if present, have been found to influence the patient's life expectancy. Each item has a weight in the index, which can be 1, 2, 3 and 6. The age ranges are also scored from 0 to 5.
HADS questionnaire (Annex 11) | day 9
  It is a scale that evaluates patients' anxiety and depression status (Zigmond & Snaith, 1983). One of its main attractions is that it suppresses somatic symptoms so that it can be evaluated independently of the underlying somatic disease. It consists of 14 items on a Likert scale of 4 points (range 0 - 3) to assess anxiety and depression (7 items for each). The total score is the sum of the 14 items (range 0 - 42), and for each subscale the score is the sum of the 7 items (range 0 - 21). It is considered that between 0 and 7 it does not indicate case, between 8 and 10 it would be a doubtful case and the scores superior to 11 are, probably, cases in each one of the subscales.
CAT Scale (Annex 12) | day 9
  The CAT scale (Jones et al., 2009) measures the impact that COPD is having on the well-being and daily life of patients. It consists of 8 items (cough, sputum, tightness in the chest, shortness of breath climbing slopes / stairs, limitation of activity in the home, confidence to leave home, sleep and energy). Each item is valued on a scale of 6 points with different formats semantically (from 0 to 5), with a total score from 0 to 40. A score between 0-10 would be indicative of a low impact of the disease.
Modified MRC scale (Annex 13) | day 9
  The modified MRC scale (Mahler & Wells, 1988) uses a very simple grading system to obtain the degree of dyspnea of the patient. This scale does not define the sensation of drowning per se, but it shows the degree of alteration that said drowning exerts on a day-to-day basis. It consists of 5 degrees of physical activity that provokes dyspnea that ranges from 0 (no type of exercise is capable of inducing dyspnea) and 4 (dyspnea prevents the patient from leaving the house or doing activities such as dressing or grooming). A higher score would be indicative of a greater degree of functional limitation.
PROactive questionnaire (Annex 14) | day 9
  This questionnaire about physical activity is a hybrid tool that combines results perceived by patients (PRO) and given physical activity objectives that come from the accelerometer (Gimeno-Santos et al., 2015). The version for clinical visit (Clinical visit PROactive PRO) will be used, which gathers the experiences of physical activity of the patients in the last 7 days. It consists of 12 questions and 2 variables of the accelerometer (14 items in total), with options on a Likert scale of 0 to 4 points, and with a score that ranges between 0 and 56 points.
Accelerometer (Annex 15) | from day 2 to 8
  The accelerometer is a motion sensor that uses a pinzoelectric transducer to detect acceleration movements in any of the 3 space dimensions (antero-posterior, medial-lateral, and longitudinal). Continuous monitoring of the actual physical activity of each patient will be obtained through a triaxial accelerometer (Dynaport® MoveMonitor) for a week. The accelerometer will be placed on all participants on the day of the IC signature. The device will be programmed to start the measurement on the day following V0 (day 2). The patient will be instructed to carry the device 24 hours a day for the next 7 days (day 2-8).
Proof of the march (PM6M) (Annex 16) | day 9
  It is a physical activity test to evaluate the effort capacity, being very simple and easy to perform, with the use of very little equipment (Holland et al., 2014, Singh et al., 2014). In this case, the maximum distance in meters that the patient travels in 6 minutes will be evaluated. Due to the learning factor demonstrated in this test, 2 tests will be carried out and the test in which the patient reached the greatest distance will be taken into account in the analysis.
Questionnaire on motivation to perform physical activity. | day 9
  This is the translation into Spanish of the questionnaire developed by Danilack et al, 2014 It consists of 4 domains (motivation, confidence, physical environment and social support) For the general reasons of motivation and trust, the subjects were asked: In general, how motivated are you to walk every day? And How confident do you feel you can walk every day? with responses on a Likert scale from 1 to 10, where the highest scores reflect greater motivation and confidence. In addition, motivation and confidence were characterized to evaluate the reasons for walking and the confidence to exercise in different situations, including health reasons, bad weather, low energy, lack of time and fear of injury.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Morell, Study Director — Fundacio Catalana de Pneumologia
Locations (1):
- FUCAP, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Pending confirmation with sponsor